CLINICAL TRIAL: NCT02346786
Title: Epidemiology of Incidents and Accidents in Sport. Influence of Moisture.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre de Recherche Rhumatologique et Thermal (Other)
Responsible Party: Principal Investigator, FORESTIER Romain, President, Centre de Recherche Rhumatologique et Thermal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CRRhumatologique
Record Dates: First submitted 2015-01-21; First posted 2015-01-27 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Fractures; Sprain; Stress Fractures; Aches; Tendinitis
Keywords: Drinking Water; Mineral water; Sports; Accident prevention
MeSH Terms: conditions — Fractures, Bone; Sprains and Strains; Fractures, Stress; Pain; Tendinopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mineral Water (Experimental): mineral water
  Interventions: Dietary Supplement: eau minérale d'Aix-Les-Bains
- Tap Water (Active Comparator): usual water intake
  Interventions: Dietary Supplement: tap water

INTERVENTIONS:
Dietary Supplement: eau minérale d'Aix-Les-Bains — Sodium 0.44 mg Magnésium 2.25 mg Phosphore 0.003 mg Potassium 0.08 mg Calcium 8.23 mg Manganèse 0.0001 mg Fer 0.001 mg Cuivre 0.0005 mg Zinc 0.0005 mg Sélénium 1 µg Iode 0 µg
  Arms: Mineral Water
Dietary Supplement: tap water
  Arms: Tap Water

SUMMARY:
sports accidents and incidents are relatively frequent. We hypothesize that the pursuit of good hydration, including days without training or competition could prevent their occurrence

DETAILED DESCRIPTION:
Main objective: to show, among practicing sports club that regular hydration, including days without competition may prevent the occurrence of an incident or accident during sport.

Primary endpoint: number of accidents and sport incidents, - Adverse events and complications at 3 months and 6 months.

EXPERIMENTAL PLAN: randomized clinical trial of two groups of athletes:

* dismissed the first group consume water from Aix-les-Bains in quantity defined during the 6 months of the study.
* Licensees 2nd group (control group) will have a free hydration, at their convenience and habits during the 6 months of the study. They will be able, if they wish to receive water from Aix within 3 months of the study.

NATURE OF TREATMENT: daily intake of Aix 1.5l water baths according to European recommendations (1 liter for children under 16 years) POPULATION STUDIED

Features licensees:

* Licensee aged 10 to 80 years;
* Practitioners sport regularly at a health club Number of members: as this is a pilot study will enroll a maximum of volunteers in each of the two clubs, a staff of 50 athletes per group is expected.

STATISTICAL ANALYSIS The variables are described (number and frequency for categorical variables, mean, standard deviation, median and confidence interval for continuous quantitative variables). The initial comparability of the two groups will be tested.

The primary endpoint will be analyzed using a Chi-square test without continuity correction if the validity conditions are true or if otherwise by Fisher's exact test. The usual additional criteria (relative risk and 95) will be presented.

For the analysis of quantitative secondary endpoints, the Student t-test will be used. If distribution does not meet the normal distribution, the nonparametric Mann-Whitney will be used. The percentage change in the activity score between baseline and 6 months 3 months will be calculated.

The qualitative evaluation criteria will be analyzed by Chi-square test without continuity correction if the conditions of validity is checked or if otherwise by Fisher's exact test.

An analysis of variance with repeated measures (comparison Inclusion- 3 months - 6 months) will be made on the physical activity score taking into account the treatment factor and interaction repetitions X treatment.

ELIGIBILITY:
Inclusion Criteria:

* Sports practitioners aged 12 to 80 years;
* Enrolled in one of two clubs participating in the study

Exclusion Criteria:

* Pregnant or breastfeeding.
* Major Licensee protected by law or deprived of liberty by administrative and judicial decisions;
* Licensee with an contra-indication for drinking water of Aix (anuric renal failure for example)
* Having dismissed contra-indication for sport practice (unlikely event, regulation of clubs requiring a medical certificate)

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-11 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
number of incidents and accidents in sport practice | 6 months

SECONDARY OUTCOMES:
estimated level of physical activity | 6 month
Warm-up time | 6 months
weigh | 6 months